CLINICAL TRIAL: NCT07296523
Title: Expert Consensus on the Use of Isotretinoin in Acne Vulgaris: A Delphi Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Isotretinoin-ACNE-VenusRC
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Isotretinoin; Isotretinoin Adverse Reaction; Acne
Keywords: Acne; Consensus; Isotretinoin; Delphi
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: A cohort of dermatology and aesthetic medicine experts participating in a Modified Delphi process to develop consensus recommendations on Isotretinoin in Acne Vulgaris.

SUMMARY:
This study is a Delphi-based expert consensus project designed to establish evidence-informed, practical recommendations for the use of isotretinoin in acne vulgaris. Despite isotretinoin being the most effective therapy for severe and refractory acne, variations persist in its indications, dosing strategies, monitoring protocols, and safety counseling.

DETAILED DESCRIPTION:
This study is a non-interventional, methodological expert consensus project that employs a modified Delphi technique to develop standardized, evidence-informed recommendations for the use of isotretinoin in the management of acne vulgaris. Although isotretinoin is widely recognized as the most effective systemic therapy for severe and treatment-resistant acne, considerable variability exists in clinical practice regarding its indications, dosing strategies, treatment duration, laboratory monitoring, pregnancy-prevention measures, and long-term maintenance. These variations reflect differences in training, regional practice patterns, and evolving evidence.

The Delphi method was selected to achieve structured consensus while minimizing the influence of dominant individuals and allowing anonymous, iterative feedback. A steering committee will first conduct a comprehensive literature review and draft a series of clear, clinically relevant statements addressing key domains of isotretinoin use. These domains will include patient selection (severity, age, psychosocial impact), baseline evaluation, dosing approaches (standard-dose, low-dose, and flexible regimens), cumulative dose considerations, treatment duration, management of adverse effects, laboratory and clinical monitoring, mental health considerations, pregnancy-prevention strategies, relapse risk, retreatment, and maintenance therapy.

A panel of expert dermatologists with demonstrated clinical experience in acne management and isotretinoin prescribing will be invited to participate. Panelists will independently rate their level of agreement with each statement using a structured Likert scale during successive Delphi rounds. After each round, responses will be analyzed quantitatively, and anonymized feedback will be provided to participants. Statements not reaching predefined consensus thresholds will be revised based on panel input and re-evaluated in subsequent rounds until consensus or stability of responses is achieved.

The final output of this study will consist of consensus-based recommendations reflecting areas of strong agreement as well as identified areas of uncertainty or disagreement. These recommendations aim to support dermatologists in making patient-centered, safe, and effective decisions regarding isotretinoin therapy, promote consistency in clinical practice, and serve as a foundation for future guidelines and research initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified or equivalent dermatologist, Minimum of 5 years of post-certification clinical experience in the management of acne vulgaris, Regular prescribing experience with oral isotretinoin in routine clinical practice, Willingness to participate in all Delphi rounds.

Exclusion Criteria:

* Inability or unwillingness to complete Delphi rounds.• Lack of clinical experience with isotretinoin.• Industry representatives without direct clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target population:
  A purposive sample of experienced clinical dermatologists who actively manage acne and regularly prescribe oral isotretinoin. The panel will include clinicians with diverse practice settings and geographic representation relevant to the study scope.
  Panel size and rationale:
  Target enrolment: 20-35 experts.
  Rationale: this size balances breadth of opinion and feasibility for iterative Delphi rounds; it is large enough to capture diverse viewpoints yet small enough to allow meaningful, anonymized feedback and analysis.
  Minimum required for analysis: 15 panelists
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 6-12 weeks
  Level of expert consensus on key clinical statements regarding isotretinoin use in acne vulgaris, measured by the proportion of panelists achieving the predefined agreement threshold (e.g., ≥70-80% agreement) for each statement across Delphi rounds.

SECONDARY OUTCOMES:
Secondary Outcome | 6-8 weeks
  Consensus on indications for isotretinoin therapy, including severity thresholds, risk of scarring, psychosocial impact, and treatment resistance.
  Consensus on dosing strategies, including initial dosing, dose escalation, low-dose regimens, cumulative dose targets, and treatment duration.
  Consensus on laboratory and clinical monitoring protocols, including baseline and follow-up testing frequency.
  Consensus on pregnancy-prevention measures and counseling practices for females of childbearing potential.
  Consensus on management of adverse effects, including mucocutaneous, psychiatric, musculoskeletal, and metabolic side effects.
  Consensus on relapse prevention and retreatment strategies, including maintenance therapy and criteria for repeat courses.
  Identification of areas of disagreement or uncertainty where consensus is not achieved, highlighting priorities for future research.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged